CLINICAL TRIAL: NCT07162558
Title: The Effect of Child-centered Empowerment on Lifestyle of Leukemia Patients
Acronym: lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Pouran Varvani Farahani, PhD in Pediatric Nursing, Department of Nursing, Faculty of Health Science, Cyprus International University,, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PVF2025CAM004
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Leukemia Acute Lymphoid Leukemia (ALL); Lifestyle Intervention for at Least 1 Month
Keywords: Empowerment Model; Quality of Life; Pediatric Nursing; Children
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Participants in this clinical trial were randomly assigned to one of two groups: an experimental group receiving the child-centered empowerment intervention and a control group receiving routine pediatric oncology care. Both groups were followed in parallel throughout the study duration.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double-Blind (Investigator, Outcomes Assessor):
  To minimize bias, a double-blind approach was employed. The researcher responsible for data collection was unaware of the group assignments, and the statistician analyzing the results was also blinded to the allocation. The data were processed under masked labels (x1 and x2) to preserve objectivity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child-Centered Empowerment (Experimental): Behavioral: Child-Centered Empowerment Intervention
  Participants in this group receive the child-centered empowerment program, a structured behavioral intervention designed to enhance coping skills, promote self-efficacy, and improve lifestyle in children with leukemia. The program is based on four dimensions of empowerment:
  Perceived Threat: Increasing awareness of illness, its complications, and the treatment process through group discussions.
  Self-Efficacy: Practicing problem-solving and self-management techniques to strengthen self-belief, self-control, and confidence in handling illness-related challenges.
  Educational Participation: Children receive educational cards at the end of each session and are encouraged to share the learned content with family members to reinforce responsibility and engagement.
  Evaluation: Continuous follow-up and assessment of learning after each session to ensure understanding and active participation.
  Interventions: Behavioral: Child-Centered Empowerment Intervention
- Routine Care (No Intervention): Participants in this group continue with their usual oncology care and do not receive any additional empowerment training. Routine medical and nursing care is delivered according to standard clinical practice without structured behavioral interventions

INTERVENTIONS:
Behavioral: Child-Centered Empowerment Intervention — Participants in this group receive the child-centered empowerment program, a structured behavioral intervention designed to enhance coping skills, promote self-efficacy, and improve lifestyle in children with leukemia. The program is based on four dimensions of empowerment:
  Perceived Threat: Increasing awareness of illness, its complications, and the treatment process through group discussions.
  Self-Efficacy: Practicing problem-solving and self-management techniques to strengthen self-belief, self-control, and confidence in handling illness-related challenges.
  Educational Participation: Children receive educational cards at the end of each session and are encouraged to share the learned content with family members to reinforce responsibility and engagement.
  Evaluation: Continuous follow-up and assessment of learning after each session to ensure understanding and active participation.
  Arms: Child-Centered Empowerment

SUMMARY:
This randomized clinical trial aimed to evaluate the effectiveness of a child-centered empowerment model in improving the lifestyle of children with leukemia. The study focused on whether structured empowerment interventions could significantly enhance daily habits and overall well-being in pediatric oncology patients. The main research questions were:

Does the child-centered empowerment model improve the lifestyle of children with leukemia? Can this complementary and non-invasive method be considered a viable approach for supporting pediatric care?

Participants (N = 46) aged 7-13 years were randomly assigned to either the intervention group, which received empowerment training in four dimensions (perceived threat, self-efficacy, educational participation, and evaluation), or the control group, which received routine care. Pre- and post-intervention assessments were conducted using a validated lifestyle questionnaire measuring nutrition, sleep, physical activity, physical health, and stress.

DETAILED DESCRIPTION:
Study Title:

The Effect of Child-Centered Empowerment on the Lifestyle of Children with Leukemia

Study Purpose:

The aim of this study was to investigate the efficacy of a child-centered empowerment model in improving the lifestyle of pediatric patients with leukemia. The intervention was designed to strengthen coping abilities, promote healthier daily habits, and enhance overall well-being, in line with holistic and family-centered nursing principles. The study was conducted as a double-blind randomized clinical trial.

Sample Size Determination:

The statistical population of this study included school-aged children (7-13 years) diagnosed with leukemia and admitted to a pediatric oncology clinic in Tehran. A total of 46 eligible children who met the inclusion criteria were enrolled using purposive sampling. Participants were randomly assigned into experimental (n = 23) and control groups (n = 23).

Sample size was determined using the mean comparison formula based on a similar study (Shoghi et al., 2019), with Type I error set at 0.05 and power at 80%. The required sample size was calculated as 19 per group, which was increased to 23 per group to account for an anticipated 20% dropout rate.

To minimize bias, a double-blind design was used. The researcher responsible for data collection was unaware of group allocations, and the statistician analyzing the data processed them under masked labels (x1 and x2).

Tools of Data Collection:

A) Demographic questionnaire: Collected background information including age, gender, weight, height, knowledge of illness, and place of living.

B) Lifestyle questionnaire: A validated 38-item tool assessing five domains-nutrition, sleep, physical activity, physical health, and stress. Each item was rated on a 4-point Likert scale ("often" to "never"), with total scores ranging from 38 to 114, categorized as unfavorable (38-63), average (64-88), and favorable (89-114). Validity and reliability were confirmed in prior studies (Farahani et al., 2018).

C) Pre- and post-intervention lifestyle assessment: Completed by all participants before and one month after the intervention period.

Intervention:

Experimental Group:

Children and their families participated in a structured child-centered empowerment program consisting of five sessions (30 minutes each) delivered by a trained pediatric nursing expert. The intervention included four dimensions:

Perceived Threat: Increasing awareness of the illness, complications, and treatment process through group discussions.

Self-Efficacy: Practicing problem-solving and self-management techniques to strengthen self-belief and self-control.

Educational Participation: Children were provided with educational cards to share learned content with family members, reinforcing knowledge and responsibility.

Evaluation: Ongoing assessment of understanding and active involvement through follow-up questions after each session.

Instructional materials were also shared via social media (WhatsApp) to enhance family engagement.

Control Group:

Children in the control group received routine care only, with no empowerment training.

Implementation Phase:

The study was conducted in the pediatric oncology clinic in Tehran. After recruitment, children were randomly allocated into intervention or control groups based on admission order (even-numbered admissions to intervention, odd-numbered to control). All participants completed demographic and lifestyle questionnaires before the intervention, and lifestyle reassessment was conducted one month after program completion.

Ethics approval The research received ethical clearance from the Near East University Ethics Review Board with the approval number NUE/2023/117-1776. The initiative closely followed the ethical standards established by the Council of Ethics and was carried out in complete accordance with the principles outlined in the Declaration of Helsinki (1964).

Statistical Analysis:

All data were analyzed using SPSS version 25. The Kolmogorov-Smirnov test was applied to check data normality. Descriptive statistics (mean, standard deviation, and frequencies) were used for demographic data. Inferential statistics included:

Paired t-test to compare pre- and post-intervention scores within each group Independent t-test to compare differences between experimental and control groups Chi-square test to analyze categorical variables A significance level of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Children aged 7-13 years diagnosed with leukemia and admitted to the pediatric oncology clinic.

Children and parents willing to participate in the study and provide written informed consent (parents) and assent (children).

No reported history of specific mental disorders as declared by parents.

Exclusion Criteria:

Inconsistent participation in empowerment sessions (e.g., missing scheduled intervention sessions).

Withdrawal from the study by the child or family at any time. Any condition preventing the child from completing questionnaires or participating in group discussions.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Lifestyle Scores | Lifestyle scores are measured at two time points - baseline (before the intervention) and one month after completion of the empowerment program
  The primary outcome measure evaluates changes in the lifestyle of children with leukemia. Lifestyle is assessed using a validated lifestyle questionnaire covering five domains: nutrition, sleep, physical activity, physical health, and stress. The tool includes 38 items rated on a 4-point Likert scale ("often" to "never"), with higher scores indicating a more favorable lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Pouran Varvani Farahani, PhD, Principal Investigator — Study Principal Investigator PhD in Pediatric Nursing, Department of Nursing, Faculty of Health Science, Cyprus International University
Locations (1):
- Near East University, Nicosia, KKTC (Turkish Republic of Northern Cyprus), Cyprus

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers